CLINICAL TRIAL: NCT01713647
Title: Comparative, Randomized,, Single Dose, Open-label, Crossover Bioequivalence Study of LOSANET AM PLUS 10mg/100mg/12.5 mg Tablets (One Tablet) of (PHARMALINE, Lebanon) Versus NORVASC 10mg Tablets (One Tablet) of (Pfizer Canada Inc., Kirkland (Quebec)) and HYZAAR 100mg/12.5 Tablets (One Tablet) of (Merck Sharp & Dohme, Quimica de Puerto Rico, Inc, Road 2 Km. 60.3, Sabana Hoyos, Arecibo, PR 00688 for Merck Sharp & Dohme B.V. Haarlem, The Netherlands) in Healthy Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Amlodipine / Losartan/ Hydrochlorothiazide of PHARMALINE, Lebanon Under Fastion Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmaceutical Research Unit, Jordan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AMLH423/PRO-00
Record Dates: First submitted 2012-10-16; First posted 2012-10-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2012-10

CONDITIONS: Fasting
Keywords: Bio-equivalence, crossover
MeSH Terms: conditions — Fasting | interventions — Losartan; Hydrochlorothiazide

ARMS (2):
- LOSANET AM PLUS (10/100/12.5 mg) of PHARMALINE, Lebanon (Experimental): Subjects will be fasted overnight and receive one tablet by mouth in accordance with randomization table, and blood samples will be taken at specified intervals over 3 days
  intervention: Drug: LOSANET AM PLUS Amlodipine/ Losartan/Hydrochlorothiazide Other Name: NA
  Interventions: Drug: Amlodipin, losartan, HCTZ
- NORVASC & HYZAAR (100/12.5 mg) (Active Comparator): Subjects will be fasted overnight and receive one tablet of Norvasc &HYZAAR by mouth in accordance with randomization table, and blood samples will be taken over 3 days
  intervention: Drug: LOSANET AM PLUS Amlodipine/ Losartan/Hydrochlorothiazide Other Name: NA
  Interventions: Drug: Amlodipin, losartan, HCTZ

INTERVENTIONS:
Drug: Amlodipin, losartan, HCTZ
  Other Names: LOSANET AM PLUS

SUMMARY:
To assess the bioequivalence of the investigational TEST product with the marketed REFERENCE products by measurement of Plasma concentrations of Amlodipine ,Losartan, Carboxylic acid losartan metabolite & Hydrochlorothiazide in plasma and calculation of the bioequivalence parameters from those measurements followed by ANOVA and 90% confidence interval statistical evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects.
2. Ethnic Group: Arab & Mediterranean
3. Race: Mixed skin (white & black skin people).
4. Age 18-50 years
5. Body-mass index 18.5 to 30.0 kg/m2 inclusive (minimum of 50 kg weight).
6. Subject is available for the whole study period and gave written informed consent
7. Physical examination within normal ranges
8. All laboratory screening results within the normal range, or being assessed as clinically non-significant by the attending physician
9. Vital signs within normal ranges.
10. Kidney function test, Liver function test should be within normal ranges.
11. Pre dosing blood pressure more than 110/70 mmHg.

Exclusion Criteria:

1. Women of childbearing potential, pregnant and lactating women.
2. Ethnic Group (Non- Arab &/ or Non- Mediterranean)
3. History of severe allergy or allergic reactions to study drug or related drugs or heparin
4. Known history or presence of food allergies, or any surgical or medical condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
5. History of serious illness that can impact fate of drugs
6. Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeletal, neurological, hematological, liver or kidney disease, unless judged not clinically significant by the Principal Investigator, or medical designate
7. Clinically significant illness 4 weeks before study Period I
8. Serious mental disease, drug, alcohol, solvents or caffeine abuse, smoking.
9. Regular use of medication
10. Having taken medication that could affect the investigated drug product: a) Regular consumption of drugs during the two weeks prior to study initiation day, b) consumption of enzyme stimulating or inhibiting drugs (e.g. Barbiturates, Carbamazepine, Phenytoin, Amphetamine, benzodiazepine, cannabinoid, cocaine, opiates, phencyclidine, and methadone) during one month before the study initiation
11. Presence of any significant physical or organ abnormality
12. Donation of 1) at least 400 ml of blood within 60 days, or 2) more than 150 ml of blood within 30 days, or 3) more than 100 ml blood plasma or platelets within 14 days before study Period I
13. Participation in another bioequivalence study within 80 days prior to the start of this study Period I
14. Following a special diet (e.g. vegetarian) or dieting one month before the study initiation.
15. Prior history of hypersensitivity to Amlodipine besylate, Losartan Potassium & Hydrochlorothiazide.
16. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration
17. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
18. Exhausting physical exercise in the last 48 hours (e.g. weight lifting) or any recent significant change in dietary or exercise habits.
19. Any significant clinical abnormality including HBsAg, HCV, and HIV
20. Abnormal vital signs.
21. Abnormal Kidney or Liver function tests.
22. Vomiting, Diarrhea.
23. Pre dosing blood pressure less than 110/70 mmHg
24. Positive test for elicit drugs and alcohol prior to dosing in each period.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To assess the bioequivalence of Test oral formulation of LOSANET AM PLUS versus References NORVASC and HYZAAR. | 9 weeks
  To assess the bioequivalence of the investigational TEST product with the marketed REFERENCE products by measurement of Plasma concentrations of Amlodipine ,Losartan, Carboxylic acid losartan metabolite & Hydrochlorothiazide in plasma and calculation of the bioequivalence parameters from those measurements followed by ANOVA and 90% confidence interval statistical evaluation.
  Cmax Ratio: Scaled average bioequivalence will be performed. Bioequivalence limits will be defined and widened according to the variance of σw2 within subject variability for the reference based on Amlodipine, Losartan, & Hydrochlorothiazide
  AUC Ratio: The 90% confidence interval for this measure lies within an acceptance range of 80.00% - 125.00% based on Losartan, & Hydrochlorothiazide
  AUC0-72 Ratio: The 90% confidence interval for this measure lies within an acceptance range of 80.00 - 125.00 % based on Amlodipine
  Carboxylic acid Losartan metabolite will be considered as supportive data

CONTACTS AND LOCATIONS:
Overall Officials: Rana .T Bustami, Phd.pharmacy, Principal Investigator — PRU
Locations (1):
- Pharmaceutical research unit, Amman, Amman Governorate, Jordan